CLINICAL TRIAL: NCT07294430
Title: Antibody-based PET Imaging and Treatment Response in Breast Cancer Treated With an Antibody-drug Conjugate According to Current Standard Indications.
Brief Title: Antibody-based PET Imaging and Treatment Response in Breast Cancer Treated With an Antibody-drug Conjugate.
Acronym: OASISImmunoPET
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UC-TRA-2521; 2025-524369-26-00 (Other: EU)
Record Dates: First submitted 2025-11-25; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Locally Advanced or Metastatic Breast Cancer
Keywords: Advanced molecular imaging; ADC; Response
MeSH Terms: conditions — Breast Neoplasms | interventions — Chromatin Immunoprecipitation Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Locally advanced or metastatic breast cancer treated with Trastuzumab deruxtecan (T-DXd) (Experimental): Experimental advanced molecular imaging (ImmunoPET) combining the high sensitivity and resolution of positron emission tomography (PET) with the specificity of ADC target specific monoclonal antibodies.
  Interventions: Procedure: Immuno-PET

INTERVENTIONS:
Procedure: Immuno-PET — Realization of an advanced molecular imaging exam to visualize the T-DXd target (HER2) expression throughout the body, at baseline and at treatment discontinuation. This procedure relies on the administration to the patient of a radioactive tracer [89Zr]-anti-HER2.
  This experimental imaging is associated to standard FDG-PET scans for tumor assessment.

SUMMARY:
OASIS-ImmunoPET is a monocentric pilot study evaluating antibody imaging to predict response to antibody-drug conjugate (ADC), an innovative cancer targeted therapy, and potentially replace tumor biopsy. It is addressed to patients with locally advanced or metastatic breast cancer who are eligible to receive the ADC Trastuzumab deruxtecan (T-DXd) according to local approval, and who are already enrolled in OASIS study (NCT pending).

DETAILED DESCRIPTION:
Antibody-drug conjugates (ADCs) have emerged as a transformative class of cancer targeted therapies, combining the specificity of monoclonal antibodies with the potency of cytotoxic payloads. This dual mechanism allows ADCs to selectively target tumor cells while minimizing systemic toxicity, thereby offering a more refined approach compared to conventional chemotherapy.

ADCs are made of 3 components: a monoclonal antibody specifically targeting tumor cells, a highly potent cytotoxic payload, and a special linker that connects the antibody to the drug. Their multi-step mode of action implies that ADC activity relies on multiple factors, such as target distribution, target density, internalization capability, linker cleavage, payload sensitivity and tumor-microenvironment modulation.

Over the past decade, ADCs have demonstrated significant improvements in survival for patients with various solid tumors and hematological malignancies. Despite these advancements, resistance to ADCs remains a major clinical challenge. Most patients who initially respond to ADC therapy eventually develop resistance, leading to disease progression. The mechanisms underlying ADC resistance are complex and poorly understood, involving tumor heterogeneity, drug metabolism, immune evasion, and alterations in target antigen expression.

Currently, no validated predictive biomarkers exist to guide ADC selection, treatment sequencing, or resistance monitoring. As a result, clinicians lack reliable tools to personalize ADC therapy, limiting the ability to optimize patient outcomes. A deeper understanding of ADC response and resistance mechanisms is urgently needed to define and adopt optimal companion diagnostics for currently approved and forthcoming ADCs and to obtain decision support tools for selecting the optimal ADC for each patient.

The protocol OASIS (NCT pending) aims to define optimal assays for predicting resistance to several approved ADCs in patients treated according to standard indications. The OASIS-ImmunoPET protocol will explore the potential contribution of advanced molecular imaging to identify response to treatment in patients enrolled in the OASIS study.

The advent of ImmunoPET combines the high sensitivity and resolution of positron emission tomography (PET) with the specificity of monoclonal antibodies (mAb) or mAb-associated fragments used as radiotracers and as such provides a comprehensive characterization of the target distribution and the target engagement over the whole-body tumor burden labeling. ⁸⁹Zr is by far the most frequently used positron-emitting nuclide for antibody.

Gebhart et al. (2016) showed the value of adding [⁸⁹Zr]-Trastuzumab PET imaging to biopsies for the assessment of intrapatient tumor heterogeneity and for prediction of the treatment outcome in HER2-positive breast cancer patients treated with Trastuzumab emtansine (T-DM1).

This OASIS-ImmunoPET study is considered a pilot sub-study of OASIS and is designed to evaluate the association between [⁸⁹Zr]-Trastuzumab PET and response in patients with HER2-positive and HER2-low breast cancer treated with T-DXd, an ADC that was developed to target HER2-expressing cancers. We aim to explore whether resistance to T-DXd is dependent on target antigen loss or heterogeneity across tumor sites and whether there is a correlation between HER2 expression level on the tumor biopsy as determined by immunohistochemistry (IHC) and HER2 PET to understand whether Ab-radiolabelled PET scan can be used as a surrogate of tumor biopsy or treatment outcome.

Both [⁸⁹Zr]-Trastuzumab PET imaging and control FDG-PET imaging will be performed at two time points: at Baseline and at End of treatment (i.e. discontinuation for any reason). Additional control FDG-PET alone will be performed just before cycle 2 (for evaluation early response), and then every 3 cycles according to standard routine.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed a written informed consent prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent;
2. Patients enrolled in the prospective cohort of the OASIS study;
3. Patient with locally advanced or metastatic breast cancer eligible to receive T-DXd as part of their standard care;
4. At baseline imaging at least two "target" lesions fulfilling the following criteria: (1) anatomically transaxial diameter ≥ 1.5 cm and measurable per RECIST1.1. and (2) metabolically assessable with a maximum standard uptake value corrected for lean body mass (SUVmax) ≥ 1.5 x SUVmean + 2 standard deviations (SD) of the liver measured in a 3-cm-diameter spherical volume of interest (VOI) in normal liver parenchyma;
5. Patients must be willing and able to comply with the protocol for the duration of the trial;

Exclusion Criteria:

1. Patients already treated with Trastuzumab deruxtecan (T-DXd);
2. Hypersensitivity at the ImmunoPET radioligands injection;
3. Patients who are claustrophobic or unable to remain still for 30 minutes;
4. Female participant who is pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 90 days after the final administration of study treatment;
5. Person deprived of their liberty or under protective custody or guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Metabolic objective response rate | From treatment initiation to disease progression, up to 3 cycles of treatment (each cycle is 21 to 28 days).
  Metabolic objective response rate (ORR) is defined as the proportion of patients who achieved a confirmed complete metabolic response (CR) or partial metabolic response (PR) assessed by investigators according to PERCIST 1.0 after 3 cycles of treatment initiation.

SECONDARY OUTCOMES:
Metabolic objective response rate (ORR) at 6 months | From treatment initiation to disease progression, up to 6 months of treatment
  Metabolic objective response rate (ORR) is defined as the proportion of patients who achieved a confirmed complete metabolic response (CR) or partial metabolic response (PR) assessed by investigators according to PERCIST 1.0 after 6 months of treatment.
Radiological objective response rate (ORR) | From treatment initiation to objective response, up to 6 months
  Radiological ORR is defined as the proportion of patients who achieved a confirmed complete radiological response (CR) or partial radiological response (PR) assessed by investigators according to RECIST 1.1 after 3 cycles and 6 months of treatment initiation.
Progression-Free Survival (PFS) | From treatment initiation to disease progression or death, up to 3 years
  Progression-Free Survival (PFS) is defined as the time from treatment initiation to the first documented radiological or metabolic progression of disease or death, whatever the cause. Patients still alive at the cut-off time without documented progression (including lost to follow-up) will be censored at the time of the latest evaluable efficacy assessment.
Radiological progression-free survival (PFS) | From treatment initiation to disease progression or death, up to 3 years
  Radiological PFS defined as time from treatment initiation to the first documented radiological or progression of disease or death, whatever the cause.
Overall Survival (OS) | From treatment initiation to death from any cause, up to 5 years
  Overall Survival (OS) is defined as the time from inclusion to death due to any cause. Patients still alive at the cut-off time (including lost to follow-up) will be censored at the last known alive date.
Time to detection of brain metastases | From treatment initiation to brain metastasis onset, up to 5 years
  Time to detection of brain metastases as identified by [⁸⁹Zr]-Trastuzumab - PET vs standard modality (brain CT/MRI, patients' symptoms, clinical examen: presence of new or progressive lesions in the brain, confirmed by radiological imaging. Detection is considered the first instance in which metastases are identified through either [⁸⁹Zr]-Trastuzumab - PET or standard modality (brain CT/MRI, patients' symptoms, clinical examen).
Proportion of patients with change in the pattern from baseline to progression or end of treatment | From treatment initiation to disease progression or death, up to 3 years
  Proportion of patients with change in the pattern from baseline to progression or end of treatment. A positive pattern means that the entire or majority of the tumour load shows significant tracer uptake, whereas a negative pattern means the dominant part or all of the tumour load lacks significant tracer uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Pistilli, MD, PhD, Principal Investigator — Gustave Roussy Cancer Center

IPD SHARING:
Plan to Share IPD: No